CLINICAL TRIAL: NCT07107893
Title: Comparison of Double Lumen Tube Location Verification Techniques in Single Lung Ventilation: Auscultation, Fiberoptic Bronchoscopy, and Video Double Lumen Tube
Brief Title: Comparison of Double Lumen Tube Location Verification Techniques in Single Lung Ventilation
Status: Completed | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Arzu Fırat Durbilmez, assistant doctor of anesthesiology and reanimation, Kayseri City Hospital
Other Study IDs: 2024-KEAK-01
Record Dates: First submitted 2025-07-17; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer; Lung Diseases
Keywords: Double lumen tube with video; Single lung ventilation
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- grup I: Group with confirmed tube location by auscultation
- Grup II: Group with confirmed tube location by fiberoptic bronchoscope
- Grup III: The group in which double lumen tube with video was used
  Interventions: Device: double lumen tube with video

INTERVENTIONS:
Device: double lumen tube with video — Methods used to confirm tube placement in one-lung ventilation: auscultation, fiberoptic bronchoscopy, and video to evaluate double-lumen tube use
  Other Names: fiberoptic bronchoscope
  Groups: Grup III

SUMMARY:
The aim of this study was to compare auscultation, fiberoptic bronchoscopy (FOB) and video double lumen tube (VDLT) double lumen tube (DLT) location confirmation techniques in terms of intraoperative tube location confirmation time, number of tube dislocations, correction time of dislocations, FOB usage rates, lung deflation quality, postoperative sore throat, presence of hoarseness and cost in thoracic surgery patients undergoing one lung ventilation (OLV).

DETAILED DESCRIPTION:
The single-center, prospective and observational study included 93 patients aged 18-84 years, American Society of Anesthesiology (ASA) I-III, who were to undergo one-lung ventilation in the lateral decubitus position by thoracic surgery under elective conditions. Patients were randomized into Group I: Group with confirmed tube location by auscultation, Group II: Group with confirmed tube location by FOB and Group III: The group in which double lumen tube with video was used. Demographic data of the patients, intubation times, tube site confirmation times, number of type dislocation, dislocation correction time, number and duration of FOB use, quality of lung deflation, presence of postoperative sore throat and hoarseness were recorded. The three groups were compared in terms of cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo TAV and be placed in the lateral position.
* Patients with ASA scores of I-III.
* Patients aged 18-84.

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients with American Society of Anesthesiology (ASA) IV and above
* Patients with anticipated difficult intubation
* Patients requiring intubation with a right thoracic duct (CLT)
* Patients with more than three intubation attempts
* Patients who refuse to participate in the study
* Patients who will undergo TAV but will not be placed in the lateral position (sympathectomy)
* Patients with uncontrolled metabolic disease
* Mentally retarded patients
* Patients under 18 or over 84
* Patients with tracheal or airway abnormalities
* Pregnant or breastfeeding women

Ages: 18 Years to 84 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Ninety-three patients who would undergo thoracic surgery with single-lung ventilation at the Health Sciences University Kayseri City Training and Research Hospital Anesthesiology and Reanimation Clinic were evaluated for suitability.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
verification of tube location | during surgery
  The primary endpoint is the identification of a method that allows the quickest confirmation of double-lumen tube location after intubation and possible intraoperative location changes.

SECONDARY OUTCOMES:
evaluation of complications | during surgery
  The secondary endpoint was to determine the superiority of three methods over each other in preventing complications that may occur due to inadequate tube location confirmation.

OTHER OUTCOMES:
cost effectiveness | during surgery
  The other endpoint is to determine the superiority of the three methods over each other in terms of reducing costs.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri Şehir Hastanesi, Kayseri, Kocasinan, Turkey (Türkiye)

DOCUMENTS (3):
  • Study Protocol: RESEARCH PROTOCOL (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT07107893/Prot_000.pdf
  • Statistical Analysis Plan: STATISTICAL ANALYSIS (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT07107893/SAP_001.pdf
  • Informed Consent Form: INFORMED VOLUNTARY CONSENT FORM (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT07107893/ICF_002.pdf